CLINICAL TRIAL: NCT00001529
Title: Use of Granulocyte Colony Stimulating Factor (G-CSF) Mobilized Leukapheresis Collections From Healthy Volunteers to Develop Improved Methods of Stem Cell and Lymphocyte Selection for Allogeneic Transplantation
Brief Title: Improved Methods of Cell Selection for Bone Marrow Transplant Alternatives
Status: Recruiting | Type: Observational
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Collaborators: New York University and New York Genome Center (Unknown)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 960049; 96-H-0049
Record Dates: First submitted 1999-11-03; First posted 1999-11-04 (Estimated); Last update posted 2026-01-05 (Actual); Status verified 2025-11-06

CONDITIONS: Graft-Versus-Host Disease; Graft-versus-leukemia; Donor Apheresis
Keywords: G-CSF; Donor Apheresis; Graft Versus Host Disease; graft versus leukemia; Natural History; Normal Volunteer
MeSH Terms: conditions — Graft vs Host Disease | interventions — Granulocyte Colony-Stimulating Factor

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Group 1: Healthy volunteers
  Interventions: Drug: G-CSF

INTERVENTIONS:
Drug: G-CSF — After medical clearance, volunteers will undergo outpatient mobilization with daily subcutaneous injections of filgrastim (G-CSF). The first dose will be administered at the NIH Clinical Center, with one-hour monitoring for immediate reactions. Volunteers may either return to NIH for daily injections or self-administer at home after training.

SUMMARY:
Bone marrow transplants (BMT) are one form of treatment for disorders of the blood, including leukemia. However, because the procedure is often associated with potentially life-threatening reactions, it is usually reserved for patients with serious illnesses under the age of 60 years old.

One serious reaction complicating bone marrow transplants is referred to as graft-versus-host disease (GVHD). GVHD is a potentially fatal incompatibility reaction. The reaction is caused by antigens found on the cells of the patient that are not present on the cells of the donor. The antigens are recognized by transplanted white blood cells (lymphocytes). These lymphocytes begin attacking the recipient s cells and tissues and may lead to death.

In order to avoid GVHD, researchers have developed a technique using peripheral blood instead of bone marrow that allows transplantation of stem cells and removal of lymphocytes. Stem cells are the cells responsible for returning blood cell production to normal. Lymphocytes are the white blood cells that can cause GVHD.

The technique requires two steps. In the first step blood cells are collected from donors who have received doses of a growth factor. The growth factor (granulocyte colony stimulating factor) is designed to increase the production of donor stem cells.

In the second step white blood cell lymphocytes are removed from the collected blood, leaving only the stem cells.

The main goal of this study is to develop and improve the method of processing cells that are collected after stimulation with growth factor (G-CSF), by removing the white blood cell lymphocytes which can cause graft-versus-host disease (GVHD) while keeping the stem cells necessary for healthy blood cell building. In addition, researchers are interested in studying whether giving G-CSF has an effect on lymphocyte function, which may influence the immune reactions occurring in bone marrow transplantation.

DETAILED DESCRIPTION:
The NHLBI Stem Cell Transplantation program is exploring ways to make allogeneic transplantation safer and more widely applicable. Prior NHLBI transplant protocols have evaluated the strategy of using T cell depleted marrow transplants followed by delayed lymphocyte add-back to control or prevent GVHD while conserving useful donor immune function against residual leukemia and infectious agents. Over the past ten years, a number of increasingly efficient methods have been used to deplete T cells but retain stem cells, and we have shown the safety and utility of the delayed T cell add-back approach. We have also found a positive relationship between the administration of higher CD34+ cell doses and outcome. Investigation of highly purified grafts with the add-back of specific T cell populations is ongoing, and the ability to test new purification approaches and devices on clinical-scale PBSC products is critical to the continued development of new transplantation approaches in our program. This requires testing the approaches on G-CSF mobilized PBSCs collected by apheresis from healthy donors since this is the cell source that will be used in all clinical allogeneic transplantation protocols in our program.

Therefore, the primary intent of this protocol is to provide a mechanism for mobilizing, collecting, storing, and analyzing G-CSF mobilized apheresis samples from healthy volunteers. Cells will be used to develop a method of processing the cells that are collected after stimulation with G-CSF, by removing the lymphocytes, which can mediate GVHD while retaining the stem cells which are necessary for hematopoietic reconstitution. At the same time, we will study whether G-CSF administration has an effect on lymphocyte, function which may influence the immune reactions occurring in allogeneic bone marrow transplantation. Furthermore, the CD34+ cells collected will be a valuable resource for experimental studies of lymphocyte-stem cell interactions in our laboratory.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Healthy individual aged 18 to 60 years.
* No active infection or history of recurrent infection.
* Normal renal function: creatinine <1.5 mg/dL or estimated glomerular filtration rate (eGFR) >=60 mL/min/1.73 m^2, with no significant proteinuria.

Normal liver function: bilirubin <2.0 mg/dL (when unconjugated), transaminases <2.0x ULN in the absence of known liver disease.

Normal blood count: WBC 2,500-11,000/microliter, ANC >1,500/microliter, platelets >150,000/microliter, hemoglobin >12.0 g/dL.

* Normal cardiovascular function, no history of chest pain, myocardial infarction, peripheral vascular disease, transient ischemic attack, or stroke.
* Healthy female subjects of childbearing age should have a negative serum pregnancy test with one week of beginning G-CSF administration.
* Female subjects should not be lactating.
* Subject must be eligible for normal blood donation. He or she must be tested negative for syphilis (RPR), hepatitis B and C (HBsAg, Anti-HBc, Anti-HCV), HIV, HTLV-1, West Nile virus, T. Cruzi and Babesia test.
* Subject must be able to comprehend the investigational nature of the study and provide informed consent to participate in the protocol.
* Antecubital veins must be adequate for peripheral access during apheresis. Potential participants must be screened by an apheresis nurse to check venous access before protocol entry.

EXCLUSION CRITERIA:

* Active viral, bacterial, fungal or parasite infection.
* Female with positive pregnancy test or lactating.
* Active or moderate-to-severe autoimmune disease that is currently treated or expected to require immunosuppressive therapy. Candidates with stable, well-controlled mild autoimmune disease may be considered on a case-by-case basis.
* Active or recent malignancy within the past 5 years. Individuals with remote (>5 years) histories of low-risk malignancies in remission (e.g., localized prostate cancer) or treated basal cell carcinoma may be included.
* History of any hematologic disorders.
* History of clinically significant cardiovascular disease (e.g., symptomatic coronary artery disease, uncontrolled hypertension). Minor risk factors must be evaluated on a case-by-case basis (e.g., controlled hypertension).
* Any positive serum screening test as listed in eligibility.
* Allergy to G-CSF or bacterial E coli products.
* Administration of NSAID within. 5-7 days of starting the protocol, depending on drug half-life.
* History of G-CSF administration and leukapheresis within past 3 months.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Healthy Volunteers
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 1996-03-18 (Actual)

PRIMARY OUTCOMES:
Provide a source of primitive hematopoietic cells from mobilized blood for laboratory studies including optimization of culture and expansion, preservation techniques, gene transfer, analysis of cell surface antigens, & analysis of migra... | End of Study

SECONDARY OUTCOMES:
Use the cells to develop a reliable technique for T cell depletion of peripheral blood stem cell transplants, which conserves sufficient CD34 cells for safe engraftment while minimizing the risk of GVHD.
Study the effect of G-CSF on lymphocyte subsets and helper cytotoxic function.

CONTACTS AND LOCATIONS:
Overall Officials: Andre Larochelle, M.D., Principal Investigator — National Heart, Lung, and Blood Institute (NHLBI)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

REFERENCES:
- [Background] Goldman J. Peripheral blood stem cells for allografting. Blood. 1995 Mar 15;85(6):1413-5. No abstract available. PMID 7534129
- [Background] Grigg AP, Roberts AW, Raunow H, Houghton S, Layton JE, Boyd AW, McGrath KM, Maher D. Optimizing dose and scheduling of filgrastim (granulocyte colony-stimulating factor) for mobilization and collection of peripheral blood progenitor cells in normal volunteers. Blood. 1995 Dec 15;86(12):4437-45. PMID 8541532
- [Background] Cottler-Fox M, Cipolone K, Yu M, Berenson R, O'Shaughnessy J, Dunbar C. Positive selection of CD34+ hematopoietic cells using an immunoaffinity column results in T cell-depletion equivalent to elutriation. Exp Hematol. 1995 Apr;23(4):320-2. PMID 7534711
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_1996-H-0049.html